CLINICAL TRIAL: NCT04061525
Title: Motion and IntraCoronary Ecg Ischemia Development Study (MICE)
Acronym: MICE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University National Heart Hospital (Other)
Responsible Party: Principal Investigator, Dobrin Vassilev, Professor, Alexandrovska University Hospital
Other Study IDs: MICE-102019
Record Dates: First submitted 2019-08-15; First posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Ischaemic Heart Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with coronary bifurcation lesions: Patients from 18 to 90-years old with coronary bifurcation lesions with significant >50% diameter stenosis artery scheduled for intervention of the main vessel (Medina types: 1x1, x11, 111)
  Interventions: Procedure: Percutaneous coronary intervention with FFR measurement and intracoronary ECG registration

INTERVENTIONS:
Procedure: Percutaneous coronary intervention with FFR measurement and intracoronary ECG registration — Measurement of fractional flow reserve (FFR), registration of intracoronary ECG and radioscopic registration of wire tip movement in the main and in the side branch in the beginning, at the end and during every step of coronary bifurcation percutaneous intervention.

SUMMARY:
The concept of the "ischemic cascade" is generally accepted hypothesis, according to which whenever ischemia of the myocardium occurs there is a consequence of events, that always occur in a given order - diastolic dysfunction first, followed by systolic dysfunction, then changes on electrocardiogram (ECG) and finally chest pain sensation. The occurrence of every next stage of cascade means more severe ischemia and respectively - more severe myocardial damage. We propose that mechanical and electrical changes in the myocardium during ischemia appear simultaneously.

DETAILED DESCRIPTION:
The development of an ischemic event, whether silent or painful, represents the cumulative impact of a sequence of pathophysiologic events. Each ischemic episode is initiated by an imbalance between myocardial oxygen supply and demand that may ultimately be manifested as angina pectoris. The ischaemic cascade is the concept that progressive myocardial oxygen supply-demand mismatch causes a consistent sequence of events, starting with metabolic alterations and followed sequentially by myocardial perfusion abnormalities, wall motion abnormalities, ECG changes, and angina. This concept would suggest that investigations that detect expressions of ischaemia earlier in the cascade should be more sensitive tests of ischaemia than those that detect expressions appearing later in the cascade.Visualization of a regional decrease in the systolic movement of the endocardium and a decrease in myocardial thickening are the main principles for the diagnosis of myocardial damage. However, the concept of ischaemic cascade is entirely based on clinical observations. It is not clear, which changes (mechanical or electrical) appear first during an episode of ischemia and which are prognostically more important. The objective of this study is to compare ischemic cascade towards ischemic constellation regarding beginning, duration and sequence of the electric, kinetic and haemodynamic signs of ischemia by FFR, icECG and wall motion abnormalities sign (M-sign - deformation and shortening of the wire tip) in patients with coronary bifurcation stenosis

ELIGIBILITY:
Inclusion Criteria:

* Subject at least 18 years of age.
* Subject able to verbally confirm understandings of risks, benefits of receiving PCI for true bifurcation lesions, and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure.
* Target main branch lesion(s) located in a native coronary artery with diameter of ≥ 2.5 mm and ≤ 4.5 mm. Target side branch lesion(s) located in a native coronary artery with diameter of ≥ 2.0 mm.
* Target lesion(s) amenable for PCI with balloon angioplasty of the side branch.

Exclusion Criteria:

* Subjects with significant ST-T change (≥ 1mm).
* Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).
* Subjects who refuse to give informed consent.
* Subjects with the following angiographic characteristics: left main coronary artery stenosis, total occlusion before occurrence of SB, lesion of interest located at infarct-related artery.
* Subjects with LVEF < 30%.
* Subjects with moderate or severe degree valvular heart disease or primary cardiomyopathy.
* LBBB, RBBB, atrial fibrillation/flutter with no identifiable isoelectric line.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Significant, >50% diameter stenosis artery scheduled for intervention of the main vessel (Medina types: 1x1, x11, 111);
  * Side branch vessel at least 2.0 mm
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Side branch region ischemia | Percutaneous coronary intervention procedure time (up to 4 hours)
  Beginning, duration, sequence of the electric, kinetic and haemodynamic signs of ischemia, comparison between ischemic cascade and constellation.

SECONDARY OUTCOMES:
Target lesion revascularization | 12 months
  Any revascularization at the territory of previously intervention
Number of patients not alive | 12 months
  Number of patients not alive
Myocardial infarction after hospital discharge | 12 months
  Myocardial infarction according to universal definition of MI - CK-MB > 2xULN +/- symptoms +/- surface ECG changes in at least 2 leads
New onset angina or heart failure symptoms | 12 months
  New onset angina symptoms of at least CCS class II; New onset dyspnea at exertion or at rest

OTHER OUTCOMES:
Periprocedural myonecrosis - extent of post PCI enzyme elevation | 48 hours
  Troponin I elevation 1-3; 3-5; >5 x ULN Creatin phosphokinase MB fraction elevation 1-3; 3-5; >5 x ULN

CONTACTS AND LOCATIONS:
Overall Officials: Dobrin Vassilev, Principal Investigator — Principal Investigator
Locations (1):
- Alexandrovska University Hospital, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vassilev DI, Mileva NB, Yaneva-Sirakova T, Georgiev RS, Kassab G. Validation of Coronary Wire for the Acquisition of Intracoronary Electrocardiogram in Swine. Catheter Cardiovasc Interv. 2025 Nov;106(5):3030-3033. doi: 10.1002/ccd.70145. Epub 2025 Sep 7. PMID 40916341